CLINICAL TRIAL: NCT06073236
Title: The Use of Co-creation to Develop an Intervention to Engage Preschoolers in Healthy Movement Behaviors for Life: the Healthy Day Project.
Brief Title: A Co-creational Intervention to Engage Preschoolers in Healthy Movement Behaviors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BC-08724
Record Dates: First submitted 2022-12-20; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Health Behavior
Keywords: 24-hour movement behaviours; behavioural change intervention; preschoolers
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial (preschools are unit of randomization) with an intervention and a control including a pretest (T0), a posttest (T1) and a follow-up (T2)
Masking Description: Parents of preschoolers in the intervention region are aware that they are taking part in a health promoting intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive what came out of the co-creation sessions with preschoolers' teachers and parents.
  Interventions: Behavioral: The healthy day-project
- Control group (No Intervention): No intervention will be given in the control group, but they will receive the intervention after follow-up. Afterwards, teachers and parents can keep the intervention materials as an incentive.

INTERVENTIONS:
Behavioral: The healthy day-project — The content of the intervention will be based on what comes out of the cocreation sessions, which means that it is not yet possible to know what the intervention will exactly consist of. The idea is to compile two co-creation groups, both consisting of preschool teachers and preschoolers' parents. Within both co-creation groups, feasible and easy-to-use strategies to implement both at preschool and at home embedded within preschoolers' play-based learning will be the goal. Both co-creation groups will investigate and develop ways to incorporate play-based learning within health promotion throughout the day at home and at preschool.
  Arms: Intervention group

SUMMARY:
Previous research focusing on preschoolers' healthy behaviors looked at developing interventions for separate behaviors, such as physical activity and sedentary behavior. Currently, there is a shift in research towards focusing on an integrated approach regarding the behaviors conducted in a 24-hour day, since targeting multiple behaviors is more effective. Activities in a 24-hour day consist of physical activity, sedentary behavior and sleep. Only very few Belgian preschoolers (10%) meet the guidelines regarding a healthy 24-hour day. Therefore, interventions focusing on all three behaviors with an integrated approach are needed. Since preschool children spend most of their time at school and at home, and engage in playbased learning in those settings, this project will develop and evaluate an intervention focusing on those 24-hour behaviors both at school and at home. The aim of the intervention is to increase the percentage of preschoolers that comply with the guidelines regarding a 24-hour day. Within the project, we will work closely together with both preschoolers' teachers and parents to develop and create the intervention, framed within the Intervention Mapping protocol. The intervention will be evaluated through a cluster randomized controlled trial, using a pretest, posttest and follow-up. Preschoolers' physical activity, sedentary behavior and sleep will be measured using an objective measurement device (accelerometer).

DETAILED DESCRIPTION:
Research has shown that sufficient physical activity, limiting sedentary behavior (i.e. sitting or lying down), and adequate sleep yield health benefits in preschoolers. This resulted in separate health guidelines for preschoolers that recommended 180 minutes of daily physical activity, spending no more than 1 hour per day sedentary in front of a screen, and sleeping at least 10h-13h per day (naps during the day included). However, research has shown that these 3 behaviors are related to each other within the time frame of a 24-hour day.

A day consists of exactly 24 hours that are filled with activities that can be categorized as physical activity, sedentary behavior or sleep. This implies that a change in one of these behaviors (e.g. more physical activity) causes a change in the time that can be spent on (one of) the other two behaviors (e.g. less sedentary and/or less sleep). Recent research has shown additional health benefits when preschoolers meet more than one of the above guidelines. For example, more positive health effects are obtained when sedentary behavior is reduced and replaced by more physical activity while maintaining the hours of sleep per day. These findings resulted in the integrated 24-hour guidelines for physical activity behavior distributed by the World Health Organization in 2019. According to these guidelines, a healthy day for preschoolers consists of (1) at least 180 minutes of physical activity, 60 minutes of which are at moderate to high intensity, (2) a maximum of 1 hour of sedentary screen time, and (3) 10 to 13 hours of good quality sleep. The greatest health effect is obtained when children meet all three guidelines.

Evidence showed that only 1 in 10 Belgian preschoolers meet the 24-hour guidelines for physical activity. Therefore, there is currently a need to develop interventions that focus on the 3 behaviors simultaneously. In the past, interventions mainly focused on one or two of these behaviors separately and never aimed for an optimal combination of these 3 behaviors. The present project will therefore develop, implement and evaluate an intervention to promote these 3 behaviors through the home and school environment. The goal of the intervention is to increase the number of preschoolers who achieve the integrated 24-hour movement behavior guidelines per day. The intervention will be developed based on the Intervention Mapping protocol, a widely used protocol to develop evidence based behavior change interventions. To increase the chance of developing a successful intervention, the intervention will be developed by using a co-creational approach. This is a specific form of collaboration where stakeholders are involved in the developmental process and the end result of the intervention. Important stakeholders for the development of preschoolers in this project are teachers and parents. Co-creation can only be successful if there is equality between the participants, reciprocity and if is conducted within an atmosphere of openness and confidence. In order for these conditions to be met, the co-creation process will be supervised by a researcher. Two co-creation groups will be formed that include both parents and teachers. Both groups will be composed of 3 to 4 preschool teachers and 3 to 4 parents of 3- to 5-year-old preschoolers. The co-creation groups will go through the first four steps of the Intervention Mapping protocol together with the researcher. The results of the co-creation will be compared after each session with the goal of reaching a consensus on the final intervention in both groups at the end of the process. The intervention will be composed of easily usable and achievable intervention strategies (e.g. storytelling, games,...) aimed at the game-based learning of preschoolers in the home and school environments.

The second objective of this research project is the evaluation of this newly developed, theory-based intervention. The intervention will be tested via a cluster randomized controlled trial (RCT) design (as preschools will be the unit of randomization), including an intervention and control group. The evaluation of the intervention will consist of an effect evaluation evaluation. We hypothesize that the intervention will lead to a higher percentage of preschool children complying with these guidelines. The design of the RCT (pretest-posttest-follow-up, intervention and control group) will allow us to measure the evolution over time as a result of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* preschoolers aged 3-5 years attending participating preschools

Exclusion Criteria:

* none

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Compliance with 24-hour movement behaviour guidelines | Pretest (before intervention)
  Compliance with 24-hour movement behaviour guidelines
Compliance with 24-hour movement behaviour guidelines | posttest (after intervention = 6 months after pretest)
  Compliance with 24-hour movement behaviour guidelines
Compliance with 24-hour movement behaviour guidelines | Follow-up (6 months after posttest)
  Compliance with 24-hour movement behaviour guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Marieke De Craemer, PhD, Study Chair — University Ghent
Locations (1):
- Ghent University, Department of Rehabilitation Sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No